CLINICAL TRIAL: NCT03749057
Title: Early Rivaroxaban for Acute Ischemic Stroke or TIA Patients With Atrial Fibrillation: a Prospective, Multicenter, Cohort Study
Brief Title: Early Rivaroxaban for Acute Ischemic Stroke or TIA Patients With Atrial Fibrillation
Acronym: ERSAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Department Chairman, General Hospital of Shenyang Military Region
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: k （2018）39
Record Dates: First submitted 2018-11-16; First posted 2018-11-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Infarction; TIA
Keywords: rivaroxaban
MeSH Terms: conditions — Cerebral Infarction | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rivaroxaban (Other): 15-20 mg rivaroxaban daily
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 15-20 mg daily

SUMMARY:
Anticoagulant treatment for non-valvular atrial fibrillation (AF) associated with cerebral infarction/ TIA is one of the recognized treatment of stroke prevention. The ACC/AHA and national guidelines for the management of anticoagulation recommend that most of AF patients with cerebral infarction or TIA should be administrated anticoagulant therapy within 14 days of symptom onset, while European guidelines recommend that the timing of the initiation of non-vitamin K antagonist oral anticoagulants (NOACs) for AF patients with cerebral infarction or TIA is association with stroke severity in light of the "1-3-6-12" principle. However, there are still many problems about the use of NOACs in ischemic stroke with AF. for example, it is unclear what time to begin NOACs as to difference in stroke severity, ages, comorbidity with hypertension, diabetes, heart failure, liver and kidney dysfunction and bleeding risks. Thus, the timing of the initiation of NOACs is yet to be further studied. Current urgent need is to develop a guideline-based specific regimen in which the benefit-risk factors are further balanced with a combination of NHISS, CHA2DS2-VASC and HAS-BLED score.

Rivaroxaban, a direct coagulation factor Ⅹa inhibitor, blocks the formation of the clot. ROCKET-AF study has shown that the efficacy of rivaroxaban is not inferior to that of warfarin in AF patients on stroke prevention, and rivaroxaban has a significantly decreased bleeding risk compared with warfarin. Recent study indicates that early administration with rivaroxaban for AF patients within 14 days of onset does not significantly increase hemorrhagic transformation. However, the relevant clinical data of the efficacy and safety of early initiation of rivaroxaban in AF patients with cerebral infarction or TIA are lacking in China.

Therefore, the investigators conduct a multicenter cohort study to investigate the safety of early rivaroxaban in the AF patient with cerebral infarction or TIA within 12 days of onset.

ELIGIBILITY:
Inclusion criteria:

1. Over 18 years
2. Acute cerebral infarction caused by non-valvular atrial fibrillation
3. NIHSS score ≤ 15
4. Within 12 days of onset
5. first stroke onset or past stroke without obvious neurological deficit (mRS score≤1)
6. Signed informed consent

Exclusion Criteria:

1. Hemorrhagic stroke or mixed stroke
2. Patients with valvular atrial fibrillation or non-cardiogenic cerebral infarction
3. Patients with severe infection or serious diseases
4. Gastrointestinal bleeding or major operation within 3 months
5. Planed cerebrovascular reconstruction or cardiac surgery within 3 months
6. Planed major surgery within 3 months
7. Participating in other clinical trials within 3 months
8. Unsuitable for this trial assessed by research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
incidence of intracranial hemorrhage | 7 days

SECONDARY OUTCOMES:
incidence of early neurological deterioration | 7 days
  2 or more increase in NIHSS
recurrence of stroke or other vascular events | 90 days
bleeding event | 90 days
  Any bleeding event except intracranial hemorrhage
Serious adverse events | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Chen, Doctor, Study Chair — Neurology Department
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, China